CLINICAL TRIAL: NCT04597827
Title: Metacognition in Semantic Dementia: Comparison With Alzheimer's Disease
Acronym: META-DEM
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.282; 2020-A02236-33 (Other: ID RCB)
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Semantic Dementia; Alzheimer Disease; Healthy
MeSH Terms: conditions — Frontotemporal Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Semantic dementia: Diagnosis of semantic dementia (revised criteria Moreaud et al., 2008; based on Neary et al., 1998)
  Interventions: Other: Metacognition tests
- Alzheimer's disease: NIAAA 2011 criteria
  Interventions: Other: Metacognition tests
- Control: MMSE above 27, no neurological or psychiatric disorder
  Interventions: Other: Metacognition tests

INTERVENTIONS:
Other: Metacognition tests — Test on episodic or semantic memory

SUMMARY:
This study aims at exploring patients' ability to monitor their own memory performance depending on their primary deficit and the type of memory involved in the criterion task. The goal is to evaluate if semantic dementia (SD) and Alzheimer's disease (AD) differently affect patients' awareness of their memory abilities.

DETAILED DESCRIPTION:
Patients who will give their informed non-opposition will be included. Participants will undergo 6 metacognitive tasks in which they will be tested on newly learnt information (i.e., episodic memory) or prior knowledge (i.e., semantic memory) and asked to evaluate their performance either prior or after the test. Correlation between their evaluation and their actual performance will be measured. Performance and correlations will be compared across groups.

ELIGIBILITY:
Inclusion Criteria:

* native French-speakers
* normal or corrected-to-normal vision
* for patients ONLY : doctor-approved diagnosis of semantic dementia or Alzheimer's disease
* for healthy participants ONLY: score above 27 on the MMSE
* non-opposition in participation

Exclusion Criteria:

* other neurological/ psychiatric disorder, or cognitive disorder that might affect general cognition
* drug or alcohol abuse

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer's disease will be patients at the CHU of Grenoble.
  Patients with Alzheimer's disease will be recruited in the CHU Grenoble, CHU Angers, CHU Bordeaux, CHU Colmar, CHU Lyon, CHU Rennes and CHUV Lausanne.
  Controls will be recruited via the database "Seniors pour la Science ", https://seniorspourlascience.fr/
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Metacognitive bias on the episodic predictive judgment task | End of study : around May 2022
  Metacognitive bias will be assessed by subtracting the mean proportion of the metacognitive judgments to the actual memory performance. Bias will range from -1 (underestimation) to 1 (overestimation).
Metacognitive accuracy on the episodic predictive judgment task | End of study : around May 2022
  Metacognitive accuracy will be assessed by calculating a gamma correlation for each participant. Metacognition accuracy allows to evaluate people's ability to discriminate correct responses from incorrect responses. Gamma correlation range from -1 to 1.
Metacognitive bias on the semantic predictive judgment task | End of study : around May 2022
  Metacognitive bias will be assessed by subtracting the mean proportion of the metacognitive judgments to the actual memory performance. Bias will range from -1 (underestimation) to 1 (overestimation).
Metacognitive accuracy on the semantic predictive judgment task | End of study : around May 2022
  Metacognitive accuracy will be assessed by calculating a gamma correlation for each participant. Metacognition accuracy allows to evaluate people's ability to discriminate correct responses from incorrect responses. Gamma correlation range from -1 to 1.
Metacognitive bias on episodic global judgment task | End of study : around May 2022
  Metacognitive bias will be assessed by subtracting the mean proportion of the metacognitive judgments to the actual memory performance. Bias will range from -1 (underestimation) to 1 (overestimation).
Metacognitive bias on semantic global judgment task | End of study : around May 2022
  Metacognitive bias will be assessed by subtracting the mean proportion of the metacognitive judgments to the actual memory performance. Bias will range from -1 (underestimation) to 1 (overestimation).
Metacognitive bias on the episodic retrospective judgment task | End of study : around May 2022
  Metacognitive bias will be assessed by subtracting the mean proportion of the metacognitive judgments to the actual memory performance. Bias will range from -1 (underestimation) to 1 (overestimation).
Metacognitive accuracy on the episodic retrospective judgment task | End of study : around May 2022
  Metacognitive accuracy will be assessed by calculating a gamma correlation for each participant. Metacognition accuracy allows to evaluate people's ability to discriminate correct responses from incorrect responses. Gamma correlation range from -1 to 1.
Metacognitive bias on the semantic retrospective judgment task | End of study : around May 2022
  Metacognitive bias will be assessed by subtracting the mean proportion of the metacognitive judgments to the actual memory performance. Bias will range from -1 (underestimation) to 1 (overestimation).
Metacognitive accuracy on the semantic retrospective judgment task | End of study : around May 2022
  Metacognitive accuracy will be assessed by calculating a gamma correlation for each participant. Metacognition accuracy allows to evaluate people's ability to discriminate correct responses from incorrect responses. Gamma correlation range from -1 to 1.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MOREAUD, Principal Investigator — University Hospital, Grenoble
Locations (7):
- France (6):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - Hôpital Neurologique de Lyon, Bron
  - Hôpitaux Civils Colmar, Colmar
  - Chu Grenoble Alpes, Grenoble
  - CHU Rennes, Rennes
- CHU Vaudois, Lausanne, Switzerland